CLINICAL TRIAL: NCT01551563
Title: Management of Inflammatory Bowel Disease in the Stavanger Area - a Prospective Evaluation of Standardized Treatment Regimens on Disease Outcome With Focus on Mucosal Healing and Associations to Fatigue
Brief Title: Stavanger University Hospital Inflammatory Bowel Disease Trial
Acronym: SUSI
Status: Recruiting | Type: Observational
Sponsor: Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Other Study IDs: SUSI_1
Record Dates: First submitted 2012-03-08; First posted 2012-03-12 (Estimated); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: IBD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and mucosal biopsies Fecal sampling
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
The study aims at studying the outcomes of a protocol-based handling of newly diagnosed Inflammatory bowel disease ( IBD ) patients within a defined uptake area in Norway. It is a descriptive study and no hypothesis is predefined.

Cytokine studies, QoL and fatigue assessment will be included for hypothesis-generating purposes.

DETAILED DESCRIPTION:
none considered needed

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed IBD

Exclusion Criteria:

* previous IBD with specific treatment within 10 year
* inability to consent
* inability to adhere to treatment protocol

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All newly diagnosed IBD patients (Crohns and Ulcerative colitis) within Stavanger Univ Hospital catchment area
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2012-04; Primary Completion 2026-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Clinical efficacy of IBD drug therapy | 5 years
  Endoscopic, clinical and biochemical response

SECONDARY OUTCOMES:
Fatigue in patients with coeliac disease - substudy | 1 year
  Fatigue severity and prevalence at diagnosis and after one year of gluten free diet
Fatigue in IBD | 5 years
  Fatigue severity and prevalence at diagnosis and during follow-up
IBD and the intestinal microbiome | 5 years
  Microbiome/eukaryome profiles associated with disease activity and treatment response from diagnosis and during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Tore Grimstad, PhD, Principal Investigator — Helse Stavanger HF
Locations (1):
- SUS, Stavanger, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Skjellerudsveen BM, Omdal R, Hetta AK, Kvaloy JT, Aabakken L, Skoie IM, Grimstad T. Less, but not gone-gluten-free diet effects on fatigue in celiac disease: a prospective controlled study. Front Med (Lausanne). 2023 Sep 12;10:1242512. doi: 10.3389/fmed.2023.1242512. eCollection 2023. PMID 37766922
- [Derived] Grimstad T, Skoie IM, Doerner J, Isaksen K, Karlsen L, Aabakken L, Omdal R, Putterman C. TWEAK is not elevated in patients with newly diagnosed inflammatory bowel disease. Scand J Gastroenterol. 2017 Apr;52(4):420-424. doi: 10.1080/00365521.2016.1273382. Epub 2016 Dec 31. PMID 28040992
- [Derived] Grimstad T, Norheim KB, Isaksen K, Leitao K, Hetta AK, Carlsen A, Karlsen LN, Skoie IM, Goransson L, Harboe E, Aabakken L, Omdal R. Fatigue in Newly Diagnosed Inflammatory Bowel Disease. J Crohns Colitis. 2015 Sep;9(9):725-30. doi: 10.1093/ecco-jcc/jjv091. Epub 2015 May 19. PMID 25994356